CLINICAL TRIAL: NCT07366619
Title: Diagnostics of the Anterior Cruciate Ligament (ACL) Using Magic Angle Directional Imaging (MADI)
Brief Title: Magic Angle Direction Imaging (MADI) ACL Study
Acronym: MADI
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 23CX8305; IRAS 301889 (Other: HRA)
Record Dates: First submitted 2026-01-05; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Anterior Cruciate Ligament Injuries; Meniscus Tear
Keywords: magic angle; musculoskeletal; low field; magnetic resonance imaging (MRI); knee; ACL; degenerative meniscus; patellar tendon; magic angle directional imaging (MADI); short T2; collagen fibre orientation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing clinically indicated MRI for investigation for ACL injury: Patients will be recruited from ICHT orthopaedic / sports medicine clinic who have suffered an ACL injury who have also undergone clinically indicated MRI
  Interventions: Diagnostic Test: Magnetic Resonance Imaging

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging — Patients will be scanned in a prototype MRI scanner at several orientations of the MRI magnet relative to the body.
  Other Names: Magic Angle Directional Imaging (MADI)

SUMMARY:
This study will be conducted to see if a new Magnetic Resonance Imaging (MRI) scanner could give additional information or help view the body in a different way. The new scanner may be useful to diagnose conditions affecting tissues such as ligaments, tendons and cartilage more accurately, potentially improving the quality of care by the NHS. To develop such protocols and to test the clinical capabilities of the scanner, it is necessary to evaluate the scans of healthy volunteers before recruiting patient participants.

Conventional MRI scans are unable to detect the signal from tissues such as ligaments, tendons, cartilage and cortical bone, which contain highly aligned collagen fibres and the signal decays too quickly to be captured. These tissues appear black and are only seen because of the surrounding brighter tissues. If a bright region appears, it can be a sign of an injury or disease, but it can also appear due to the Magic Angle artefacts, when the collagen fibres are at a specific angle to the main magnetic field of the MR scanner. This anomaly can make assessment of these tissues difficult. Currently the diagnostic gold standard is arthroscopy, though it is mostly undertaken therapeutically.

The method harnesses this inherent tissue property to gain information about these collagen-rich tissues in joints. Using Magic Angle Direction Imaging (MADI) it is possible to obtain detailed information about the collagen fibre structures, and this is not available using conventional MRI. MADI could be important for planning surgery, developing new tissue implants, and monitoring outcome measures.

In both standard cylindrical scanner and the conventional open scanner, it is impossible to move the magnet, nor the patient, in the required manner. This motivated the development of a novel prototype MA scanner that can move around the patient.

The aim of this study is to evaluate the ability to routinely perform in-vivo Magic Angle-MRI of collagen structures in joints based on the magic angle principle, and to assess the ability to use qualitative and quantitative assessment of the Magic Angle-MR images to distinguish between the pathologies of the soft structures imaged.

DETAILED DESCRIPTION:
STUDY DESIGN

1. Type of Study This is a pilot study investigating the potential role of MA-MRI in visualising and assessing ACL tears in the knee using a non-CE marked medical device.

   The patient study follows on from a pilot study of healthy volunteers that enabled the research team to establish the best practice and sequences for qualitative/quantitative evaluation of the knee joint.

   The MRI study protocol has been developed using healthy volunteers initially and now will be tested in patients. Methods for positioning the healthy volunteers and their limbs will now be applied to a patient cohort. The scanner is based at the Mechanical Engineering department at Imperial College London, South Kensington campus.
2. Duration It will last 36 months.
3. Number and Type of Subjects As this is a novel technique there is no data available to perform a reliable power calculation. However, similar studies to examine the efficacy of the novel MRI technique image between 20 and 30 subjects. This study will therefore recruit 20 patients. 20 healthy volunteers have previously been recruited from staff and students at Imperial College London to fine tune the methods before the patient study commences. The patient group will be recruited from ICHT sports injury/orthopaedic clinic once a diagnosis of an ACL tear has been made with conventional MRI.
4. Recruitment 20 patients will be recruited from ICHT orthopaedic / sports medicine clinic who have suffered an ACL injury who have also undergone clinically indicated MRI.

   Patients will be recruited from Charing Cross Hospital and St Mary's Hospitals. They will be identified by members of the clinical team, who are also members of the research team at ICHT. NHS systems, MDT meetings and clinics will all be used to identify appropriate patients as per the inclusion and exclusion criteria (participant entry). A poster with a QR code to contact the study coordinator should patients wish to take part in the study will be placed in the orthopaedic and sport clinic waiting room.

   The clinical team at ICHT, some of whom are also part of the research team, will identify the patients, and will inform the research team at ICHT who the potential patients are once the patients have given verbal consent to be contacted by the research team. Patients will be given details of the study (in lay language), and any queries will be addressed by the members of the research team at ICHT. Written information will also be provided in the form of a patient information sheet that accompanies an invitation letter for the study. The invitation letter will be sent if a patient contacts the team after seeing a recruitment poster, after the patient's first appointment at clinic, or later based on the waiting list for ACL surgery. A video of the scanner and its movement will also be made available to interested patients.

   The research team will then call the patients, and ensure the patient is given the Patient Information Sheet and explain the study to them. A follow up call to the patients to check if they are interested in taking part will be made. If they are interested, then this call will also involve confirming the patient's eligibility, by going through the inclusion/exclusion checklist with them, as well as the MR safety checklist. This will include asking them their height and weight to get their BMI. If they are eligible then they will be invited to take part.

   Sufficient time will be given for full consideration of participation before informed consent is obtained. They will be assured their participation is entirely voluntary and their decision will have no impact on their clinical care.

   Either written or electronic informed consent must be obtained. Patients will be contacted for a telephone conversation by members of the research team at ICHT to ask questions about the study and any concerns before they consent.

   Patients will have the option to sign an informed consent form at ICHT sites or sign e-consent on the REDCAP database before any study procedures take place, and then the complete eligibility check will be completed, by going through the inclusion/exclusion checklist with patients, including measuring height, weight and thigh circumference. The research team will also complete the MR safety checklist with the patients.

   Reasonable travel expenses will be reimbursed for participants when required, up to £20 per participant for travel to the Magic Angle scanner based at Imperial College London.
5. MRI Safety Participants will be asked to complete an MRI safety checklist to ensure that they are safe to go into an MRI scanner. Members of the study team will contact participants and confirm their eligibility according to the short MR safety check. Any red flags mean that the patient failed the eligibility criteria and cannot be included in the study. It is anticipated that they will have already been scanned on a hospital MRI system and completed the hospital MR safety form. However, before inclusion into this study the MR safety checklist will ensure there are no contraindications to MA-MRI. There is an adapted MR safety checklist which can be used to identify suitable patients at the recruitment stage.

   The research MR safety checklist is more restrictive due to the non-CE marked device and the magnetic field's ability to move around the patient. The MA-MRI scanner is low field so is unlikely to be less safe than conventional MRI, (10 times less strong). However, most safety data and recommendations are researched on horizontal field 1.5 T or 3T systems. No MR conditional active implants will be scanned on the MA-MRI system. Passive MR conditional implants may be scanned as it is unlikely that they will be inside the transmit coil (e.g., hip replacement).

   The medical physics team will review safety data for the device.

   An investigator meeting of the Trial Steering Group will be held after the first 10 patients have been scanned in order to review interim safety and efficacy of the trial.
6. Methods The MA-MRI scanner will be used for all research scans. The scanner is in the Mechanical Engineering Department at Imperial College London, South Kensington campus.

   Once participants have given either written or electronic informed consent to take part in the study, they will undergo the MA-MRI scan. Transportation will be organised for the patient to bring them to the South Kensington campus of Imperial College London where they will be met by the postdoctoral research radiographer and their consent from will be checked to verify consent. If a paper consent form was signed, a copy of the signed ICF will be taken with the patient to the Imperial College London site, for the ICL team to confirm the patient is fully consented before undergoing the MADI scan.

   The visit to the MA-MRI scanner will take about 1 ½ hours and the imaging itself will be performed over a period of about an hour. The patient will be asked to remove and lock away any jewellery or loose metal items from around the body. If needed change into MR safe clothing (scrubs) without zips or metal fastening near the joint being scanned.

   The patient will be comfortably sitting outside the MRI magnet (as opposed to conventional MRI where they will lie in a tunnel with their head at the opening). Whichever knee is being imaged either right and/or left will be positioned in the receiver coil, which is then placed between the magnetic poles on the holder to reduce any movement and ensure it is in the centre of the magnet. Padding will be applied around the thigh and calf to keep the patient comfortable. The chair will be adjusted, and leg support used to ensure the patient's comfort.

   If patients prefer (their choice) they can be given earplugs or headphones as the MRI scans can be noisy, however we have measured the scan noise to be at a similar level to speaking (60-65dB). The patient will also be provided with a panic alarm to stop scanning if they are no longer happy to continue with the study or wish to stop the scanner rotating.

   All the images will be looked over by the research team. The MA-MRI scans are not intended as a diagnostic scan, however if additional pathology is detected on the MA-MR images that were not apparent on the conventional MRI scan the Radiologist reviewing will add an addendum to the patient's record on the Imperial College Healthcare Trust's PACs record. The participants lead clinician will also be informed.

   One year (+/- one month) after the Magic Angle scan, participants will be contacted either by phone or email to identify any further pathologies that have been identified through their clinical investigations, and collection of any relevant imaging and information from their clinical notes will be collected.
7. Data Processing The raw data from the scan will be post-processed using the algorithms developed by the research team. These identify voxels in the multiple image positions that have exhibited a significant change in signal intensity which suggests they are made up from orientated collagen structures exhibiting a magic angle effect. The net collagen fibre direction of those voxels is computed then co-registered onto the initial anatomical MRI scan to aid visualisation.

   Images will be presented to and discussed with the steering group of radiologist surgeons and sports physicians for their feedback. Improvements to the imaging can be made if necessary. Quantitative measurements of width and length of tendons and ligaments and meniscus can be performed in the images.
8. Statistics and Data Analysis Radiologists will perform the visual, qualitative analysis of the MR images, and these will be assessed using descriptive purposes. These will be recorded in a record sheet. Clinical correlation with conventional MRI and operative findings (where available) will be performed.

Reviewers will be blinded to the findings of the clinical MRI studies prior to reviewing the images. Two suitably qualified reviewers within ICL and/or ICHT will review the patient images on both the conventional and the MA-MRI in different sittings, randomised order, and blinded to clinical findings.

Visual grading of the anterior cruciate ligament fibres will be assessed as per the table below. If articular cartilage and meniscus can be visualised, then a similar grading system will be used to assess the collagen fibre directions.

ACL Ligament

1. = not seen Individual 'bands' not well seen
2. = probably seen Bands seen mild-to-moderate signal with indistinct margins
3. = seen Bands well seen with mild-to-moderate signal with definitive margins
4. = readily seen Bands well seen with indistinct individual fibres
5. = well seen Circumscribed, strong signal with individual fibres seen

Visual grading of the ACL structure will be assessed as per the table below. Visual grading of patients MA-MRI to cMRI compared by statistical testing (depending on distribution) with p <0.05 indicating significant difference and the null hypothesis (no difference in grading between the MRI techniques).

Patients with ligament tear

1. = no tear 0% Individual 'bands' appear intact
2. = partial tear - low grade up to 49% PL and AM band seen with incomplete tear to one or a complete tear of one bundle
3. = partial tear - high grade over 50% Less than one bundle seen remaining
4. = complete tear 100% Complete destruction of all fibres

Arthroscopic grading Grade 1 Mild injury to the ACL such as stretching that has led to laxity and reduction of tension in the ligament.

Grade 2 Partially torn ACL Grade 3 Fully torn ACL Tibial Spine Avulsion ACL injury The ACL itself is not torn but the bony attachment of the ligament to the tibia is pulled off.

It is beyond the scope of this patient study to confirm the accuracy as no biopsy or tissue samples will be acquired for corroboration. Animal model studies alongside polarised light microscopy study will inform accuracy of the collagen fibre directions.

The recruitment target will be 20 patients with anterior cruciate ligament injury.

Data and all appropriate documentation will be stored for a minimum of 10 years after the completion of the study, including the follow-up period, as per Imperial College policies.

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 - 65 years
* selected for ligament repair surgery
* ability to give informed consent, either written or e-consent
* no contraindications to MRI
* BMI ≤ 28 or thigh circumference less than 47 cm at approximately 7.5cm above the joint line

Exclusion Criteria:

* acutely unwell or frail patients in whom extension of scanning time may not be tolerated or may delay treatment
* contraindications to MRI
* participants who are too big to be able to fit in the prototype scanner
* recent surgery to the affected joint
* severe pain
* pregnant and/or breastfeeding participants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Before a patient can enter the study, they will have undergone a clinically indicated MRI for knee pathology which diagnosed an ACL injury requiring surgery.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-29 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Reproducibility with Magic Angle MRI | Before surgery and 12 months after surgery.
  The primary outcome measures will be the reproducibility with MA-MRI in a group of patients with known ACL tears. We will use a grading system for the radiologists to assess the MA-MRI images through a) qualitative assessment to grade ACL fibres and b) quantitative assessments to distinguish between the ACL tears with a grading system for the radiologists.
  1. Visual grading of the anterior cruciate ligament fibres will be assessed (range 1-5) as follows:
     * 1 = not seen
     * 2 = probably seen
     * 3 = seen
     * 4 = readily seen
     * 5 = well seen
  2. Visual grading of the ACL structure for patients with ligament tear will be assessed as per the table below.
     * 1 = no tear 0%
     * 2 = partial tear - low grade up to 49%
     * 3 = partial tear - high grade over 50%
     * 4 = complete tear 100%

SECONDARY OUTCOMES:
Comparison of the ACLs imaged with MA-MRI against best practice | 12 months after surgery
  The secondary outcome measure will be a comparison of the ACLs (Anterior Cruciate Ligament) imaged with MA-MRI against best practice:
  1. cMR images (conventional MRI) performed pre-operatively to diagnose ACL injury taken from the imaging report and qualitative and quantitative assessment by 2 radiologists using the same scale as for MA-MR images (as defined for the Primary Outcome Measures);
  2. Arthroscopic assessment of the ACL during repair taken from surgical notes, evaluating the potential suitability of MA-MRI as a diagnostic tool for ACL injury.
  Arthroscopic grading will be as follows:
  * Grade 1 (Mild injury to the ACL such as stretching that has led to laxity and reduction of tension in the ligament)
  * Grade 2 (Partially torn ACL)
  * Grade 3 (Fully torn ACL)
  * Tibial Spine Avulsion ACL injury (The ACL itself is not torn but the bony attachment of the ligament to the tibia is pulled off)

CONTACTS AND LOCATIONS:
Overall Officials: Chinmay Gupte, PhD, Principal Investigator — Imperial College NHS Trust
Locations (2):
- United Kingdom (2):
  - Imperial College London, London
  - Imperial College NHS Trust, Department of Surgery and Cancer, London

IPD SHARING:
Plan to Share IPD: No
Data will be fully anonymised for any publication

REFERENCES:
- [Background] Valente G, Pitto L, Testi D, Seth A, Delp SL, Stagni R, Viceconti M, Taddei F. Are subject-specific musculoskeletal models robust to the uncertainties in parameter identification? PLoS One. 2014 Nov 12;9(11):e112625. doi: 10.1371/journal.pone.0112625. eCollection 2014. PMID 25390896
- [Background] Amin NH, Hussain W, Ryan J, Morrison S, Miniaci A, Jones MH. Changes Within Clinical Practice After a Randomized Controlled Trial of Knee Arthroscopy for Osteoarthritis. Orthop J Sports Med. 2017 Apr 10;5(4):2325967117698439. doi: 10.1177/2325967117698439. eCollection 2017 Apr. PMID 28451610
- [Background] Fullerton GD, Cameron IL, Ord VA. Orientation of tendons in the magnetic field and its effect on T2 relaxation times. Radiology. 1985 May;155(2):433-5. doi: 10.1148/radiology.155.2.3983395.
- [Background] Fullerton GD, Rahal A. Collagen structure: the molecular source of the tendon magic angle effect. J Magn Reson Imaging. 2007 Feb;25(2):345-61. doi: 10.1002/jmri.20808. PMID 17260393
- [Background] Bydder M, Rahal A, Fullerton GD, Bydder GM. The magic angle effect: a source of artifact, determinant of image contrast, and technique for imaging. J Magn Reson Imaging. 2007 Feb;25(2):290-300. doi: 10.1002/jmri.20850. PMID 17260400
- [Background] Du J, Pak BC, Znamirowski R, Statum S, Takahashi A, Chung CB, Bydder GM. Magic angle effect in magnetic resonance imaging of the Achilles tendon and enthesis. Magn Reson Imaging. 2009 May;27(4):557-64. doi: 10.1016/j.mri.2008.09.003. Epub 2008 Nov 20. PMID 19022600
- [Background] Szeverenyi NM, Bydder GM. Dipolar anisotropy fiber imaging in a goat knee meniscus. Magn Reson Med. 2011 Feb;65(2):463-70. doi: 10.1002/mrm.22645. Epub 2010 Oct 11. PMID 20939091
- [Background] Bydder GM. Review. The Agfa Mayneord lecture: MRI of short and ultrashort T(2) and T(2)* components of tissues, fluids and materials using clinical systems. Br J Radiol. 2011 Dec;84(1008):1067-82. doi: 10.1259/bjr/74368403. PMID 22101579
- [Background] McGinley JV, Ristic M, Young IR. A permanent MRI magnet for magic angle imaging having its field parallel to the poles. J Magn Reson. 2016 Oct;271:60-7. doi: 10.1016/j.jmr.2016.08.001. Epub 2016 Aug 8. PMID 27552556
- [Background] Jones GMC, Pitsillides AA, Meeson RL. Moving Beyond the Limits of Detection: The Past, the Present, and the Future of Diagnostic Imaging in Canine Osteoarthritis. Front Vet Sci. 2022 Mar 15;9:789898. doi: 10.3389/fvets.2022.789898. eCollection 2022. PMID 35372534
- [Background] Brujic D, Chappell KE, Ristic M. Accuracy of collagen fibre estimation under noise using directional MR imaging. Comput Med Imaging Graph. 2020 Dec;86:101796. doi: 10.1016/j.compmedimag.2020.101796. Epub 2020 Oct 9. PMID 33069034
- [Background] Chappell KE, Brujic D, Van Der Straeten C, Meeson R, Gedroyc W, McRobbie D, Ristic M. Detection of maturity and ligament injury using magic angle directional imaging. Magn Reson Med. 2019 Sep;82(3):1041-1054. doi: 10.1002/mrm.27794. Epub 2019 May 12. PMID 31081201